CLINICAL TRIAL: NCT05809700
Title: The Clinical Study of Injection of Freshly Prepared HA35 in the Treatment of Shoulder, Neck, Back, Temporal and Herpes Zoster Pain
Brief Title: Injection Therapy for Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dove Medical Press Ltd (Network)
Responsible Party: Principal Investigator, Mizhou Hui, Research fellow, The Affiliated Hospital of Qingdao University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSHN001
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HA35 local injection of pain location Group (Experimental): According to the ratio of 100 mg high molecular weight HA (sodium hyaluronate for injection, H20174089)/2000 units of hyaluronidase extracted from bovine testis (hyaluronidase for injection H31022111), high molecular weight HA injection and hyaluronidase injection were mixed at room temperature for 20 minutes.
  Interventions: Drug: Freshly manufactured 35 kDa hyaluronan fragment

INTERVENTIONS:
Drug: Freshly manufactured 35 kDa hyaluronan fragment — This mixture of high molecular weight HA and hyaluronidase containing 100 mg of HA was locally injected at the pain point or where the nerve trunk innervates the pain point. Then, the pain scale (NPRS) was used to evaluate pain, and the pain relief of patients before and after treatment was recorded.
  Each time, according to the amount of high molecular weight HA containing 100 mg HA and hyaluronidase mixture, the pain point area and pain point area of the nerve trunk innervation of the local multipoint injection. Then, the pain scale was used to evaluate pain, and the pain relief of patients before and after treatment was recorded.
  Other Names: HA35

SUMMARY:
Shoulder, neck, back and temporal pain and herpes zoster pain are neuropathic pain. Preliminary clinical studies have confirmed that injection of freshly prepared HA35 can relieve neuropathic pain. This clinical study is a prospective repeated experiments. The purpose of this study was to verify the effectiveness of HA35 injection therapy.

DETAILED DESCRIPTION:
In this study, the recombinant human hyaluronidase PH20 and neutral hyaluronidase (PH20) of bovine testicular sperm acrosomes were used to cleave macromolecular HA. Regardless of the cutting time, the HA fragment HA35, with an average molecular weight of 35 kDa, was produced (Registration number L20200708MP07707, Ministry of Health, Mongolia). Hyaluronidase is often used to improve the penetration and absorption of other injectable drugs. Hyaluronidase injection is also used off label to degrade excessive components used in cosmetic injections, such as cross-linked macromolecular HA fillers (https://www.realself.com/news/hyaluronidase-dissolve-fillers). In this study, HA35 was prepared by mixing hyaluronidase extracted from bovine testis (hyaluronidase for injection, H31022111) and HA (sodium hyaluronate for injection, H20174089) at room temperature for 20 minutes. The analgesic effect of HA35 on herpes zoster and shoulder, neck, back, and temporal pain was studied. This was a single-arm, open-label prospective clinical study in which patients were evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* The course of neck, back and temporal pain ranged from 0 to 8 months.
* The course of herpes zoster of 0-2 months.
* Adults aged 18-60 years.
* Be willing and capable of giving informed consent.
* Have a clinical diagnosis of neuropathic pain as determined by a multidisciplinary study team.
* Subject must sign the informed consent in person prior to beginning any screening procedure.

Exclusion Criteria:

* Have a persistent pain resulted from other medical conditions or unknown causes.
* Pregnant females.
* Be concomitantly participating in another clinical study.
* Have been immunocompromised.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
the Numerical Pain Rating Scale (NPRS) scores | 30 min to 3 hours
  The pain scale used is a tool that doctors use to help assess patients' pain. Each patient rated their pain on a scale of 0 to 10. A score of 0 means "no pain" and 10 means "the most painful". Statistical t-tests were used to calculate and evaluate the pain intensity, which were expressed as the mean ± standard deviation.
the General Comfort Questionnaire (GCQ) scores | 24 hours
  Using 1-4 grade scoring method, that is, 1 means ' very disagree ', 2 means ' disagree ', 3 means ' agree ', 4 means ' very agree'. The total score is less than 60 points for low comfort, 60-90 points for moderate comfort, and more than 90 points for high comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Huinuode Biotechnology Co., Ltd., Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
The data will be sent to the accepting journal study.